CLINICAL TRIAL: NCT03530696
Title: A Single Arm Phase II Study to Evaluate Efficacy of T-DM1 With Palbociclib in the Treatment of Patients With Metastatic HER2 Positive Breast Cancer
Brief Title: T-DM1 and Palbociclib for Metastatic HER2 Breast Cancer
Acronym: T-DM1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29747; T-DM1 (Other: The University of Arizona Cancer Center); Palbo T-DM1 (Other: The University of Arizona Cancer Center)
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: HER2-positive Breast Cancer; Breast Cancer; Breast Cancer Stage; Recurrent Breast Cancer; Metastatic Breast Cancer; HER2 Positive Breast Carcinoma
Keywords: Breast Cancer; HER2-positive; T-DM1; HER2-positive Breast Cancer; Recurrent Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- T-DM1 with palbociclib (Experimental): T-DM1 is given intravenously every 21 days (day 1 of each cycle) Palbociclib is administered orally on days 5-18 of each cycle
  Interventions: Drug: Palbociclib; Drug: T-DM1
- Single Agent T-DM1 (Experimental): T-DM1 is given intravenously every 21 days (day 1 of each cycle)
  Interventions: Drug: T-DM1

INTERVENTIONS:
Drug: Palbociclib — Palbociclib is to be taken orally on days 5-18 (14 days) of each cycle (each cycle length is 21 days). The starting dose will be 125mg.
  Other Names: Ibrance
  Arms: T-DM1 with palbociclib
Drug: T-DM1 — The recommended dose of T-DM1 is 3.6 mg/kg and is given as an intravenous infusion on Day 1 of every cycle (every 21 days).
  Other Names: Kadcyla

SUMMARY:
This is a single arm, phase II study to evaluate if the combination of T-DM1 with palbociclib improves progression-free survival in patients with metastatic HER2 positive breast cancer. All patients will be treated with T-DM1 with palbociclib.

DETAILED DESCRIPTION:
This is a multi-center, single arm, phase II study of T-DM1 with palbociclib in the treatment of patients with metastatic HER2-positive breast cancer.

Hypotheses: Combination of T-DM1 with palbociclib improves progression free survival

Primary objective: Progression free survival of the combination of T-DM1 with palbociclib

Secondary objectives i) Response rates ii) Overall survival

Correlative objectives i) Investigate predictive biomarkers of response in blood and archived tumor tissue ii) Investigate mechanisms of resistance for palbociclib in blood and tumor tissue

ELIGIBILITY:
Inclusion Criteria:

1. Be informed of the investigational nature of the study and all pertinent aspects of the trial
2. Sign and provide written consent in accordance with institutional and federal guidelines.
3. ECOG Performance status of 0-2
4. Recurrent or metastatic HER2-positive breast cancer (HER2 positive is defined per ASCO-CAP guidelines)
5. Adequate cardiac reserve (EF≥50%)
6. Serum creatinine ≤ 1.5 x institutional upper limit of normal (IULN), bilirubin ≤ 2.0, and an SGOT/SGPT/alkaline phosphatase ≤ 2.0 x IULN
7. Adequate bone marrow function (ANC ≥1000, Platelets ≥100,000/ml, Hemoglobin ≥10gm/dL)
8. Be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures
9. Been treated with pertuzumab previously (neoadjuvant or metastatic setting). Patients who weren't able to tolerate pertuzumab due to side effects can be eligible for study upon discussion with the study PI
10. No more than 2 lines of therapy in the metastatic disease setting

Exclusion Criteria:

1. HER2 negative tumors
2. Prior treatment with T-DM1
3. Prior treatment with CDK 4/6 inhibitors
4. Known active CNS metastases or carcinomatous meningitis. Patients with stable CNS metastases including brain metastases who have completed a course of radiotherapy are eligible for the study provided they are clinically stable. However, oral corticosteroids for control of CNS symptoms are not allowed on study
5. Known documented or suspected hypersensitivity to the components of the study drug(s) or analogs.
6. Uncontrolled systemic illness, including but not limited to ongoing or active infection
7. Symptomatic congestive heart failure, unstable angina pectoris, stroke or myocardial infarction within 3 months
8. Be pregnant or breast feeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment and must agree to use effective contraception during the period of therapy
9. Concurrent hormonal or other anti-neoplastic therapy is not allowed. Patients can receive supportive therapy like bone-directed therapy including bisphosphonates or denosumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, MD, Principal Investigator — The University of Arizona Cancer Center
Locations (16):
- United States (16):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Cedar-Sinai, Beverly Hills, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mosaic Life Care, Saint Joseph, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Roswell Park Comprehensive Cancer center, Buffalo, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - JPS Health Network, Fort Worth, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T-DM1 With Palbociclib | Single Agent T-DM1
Started | 39 | 16
Completed | 38 | 14
Not Completed | 1 | 2
Not completed — Excluded for not meeting eligibility criteria upon further review | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T-DM1 With Palbociclib | Single Agent T-DM1 | Total
Number analyzed (Participants) | 38 | 14 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Age is missing for 1 participant in the Single Agent T-DM1 arm (n=13).
  Years
    number analyzed (Participants) | 38 | 13 | 51
    (all) | 56.5 (12.6) | 57.8 (11.4) | 56.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 14 | 52
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/ethnicity is missing for 3 participants across both arms: n=36 for T-DM1 with palbociclib and n=13 for Single Agent T-DM1.
  Participants
    White: number analyzed (Participants) | 36 | 13 | 49
    White | 24 | 10 | 34
    Hispanic: number analyzed (Participants) | 36 | 13 | 49
    Hispanic | 4 | 2 | 6
    Black: number analyzed (Participants) | 36 | 13 | 49
    Black | 4 | 1 | 5
    Asian or Pacific Islander: number analyzed (Participants) | 36 | 13 | 49
    Asian or Pacific Islander | 3 | 0 | 3
    American Indian or Alaskan Native: number analyzed (Participants) | 36 | 13 | 49
    American Indian or Alaskan Native | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 14 | 52
Menopausal Status [Count of Participants; unit: Participants]
  Surgical Menopause | 3 | 1 | 4
  Pre-Menopausal | 10 | 1 | 11
  Post-Menopausal | 25 | 12 | 37
Current HER2+ Breast Cancer Diagnosis [Count of Participants; unit: Participants] — HER2 positivity is defined per American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) guidelines.
  Participants
    Metastatic | 37 | 14 | 51
    Recurrent | 1 | 0 | 1
Prior Treatment Lines in Metastatic Setting [Count of Participants; unit: Participants] — During screening, patients' medical records were reviewed to assess the number of previous treatments they received for metastatic disease.
  Participants
    0 | 13 | 4 | 17
    1 | 14 | 3 | 17
    2 | 8 | 6 | 14
    3 | 3 | 1 | 4
Pertuzumab Prior to Study [Count of Participants; unit: Participants] — The information in this table reflects the number of patients who received Pertuzumab prior to enrolling on this study (denoted by "Yes") and the number of patients who did not receive Pertuzumab prior to enrolling on this study (denoted by "No").
  Participants
    No | 11 | 4 | 15
    Yes | 27 | 10 | 37
Estrogen Receptor (ER) Status [Count of Participants; unit: Participants]
  Negative | 25 | 9 | 34
  Positive | 13 | 5 | 18
Progesterone Receptor (PR) Status [Count of Participants; unit: Participants]
  Negative | 20 | 5 | 25
  Positive | 18 | 9 | 27
Bone Metastasis [Count of Participants; unit: Participants] — Population: Bone metastasis data is missing for 1 participant in the T-DM1 with palbociclib arm (n=37).
  Participants
    No: number analyzed (Participants) | 37 | 14 | 51
    No | 22 | 9 | 31
    Yes: number analyzed (Participants) | 37 | 14 | 51
    Yes | 15 | 5 | 20
Central Nervous System (CNS) Metastases [Count of Participants; unit: Participants] — Population: CNS metastasis data is missing for 1 participant in the T-DM1 with palbociclib arm (n=37).
  Participants
    No: number analyzed (Participants) | 37 | 14 | 51
    No | 7 | 0 | 7
    Yes: number analyzed (Participants) | 37 | 14 | 51
    Yes | 30 | 14 | 44

OUTCOME MEASURES:

1. Primary Outcome: Estimate Progression-free Survival
Description: Progression Free Survival (PFS) is defined as the time from date of first treatment to the date of investigator-determined objective disease progression as defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST) 1.1 or death from any cause. Per RECIST 1.1 for target lesions: Complete Response (CR) is the disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Progressive Disease (PD) is at least a 20% increase in the sum of diameters of target lesions; Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Patients who have neither progressed nor died will be censored at the day of their last radiographic tumor assessment (if available) or date of randomization if no post initiation (that is post baseline) radiographic assessment is available.
Time Frame: Up to 4 years
Population: Number of patients included for PFS analysis:
  T-DM1 with Palbociclib Arm: n=36 T-DM1 Arm: n=11
  5 patients lack data on response because they discontinued study participation (or withdrew consent) before the first scan. Thus, the final sample size for responses is n = 47.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | T-DM1 With Palbociclib | Single Agent T-DM1
Number analyzed (Participants) | 36 | 11
Months | 16.9 [8.3 to NA] — The upper limit was not reached due to insufficient number of participants who progressed. | 8.3 [2.7 to 8.8]

2. Secondary Outcome: Number of Participants With Response
Description: Per RECIST 1.1 for target lesions: Complete Response (CR) is the disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Progressive Disease (PD) is at least a 20% increase in the sum of diameters of target lesions; Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Overall response rate (ORR) is defined as the proportion of patients with CR or PR per RECIST 1.1. Disease control rate (DCR) is defined as the proportion of patients with CR, PR or SD per RECIST 1.1. The data shown is the number of participants with ORR, DCR, CR, PR, PD, and SD.
Time Frame: Up to 4 years
Population: 5 patients lack data on response because they discontinued study participation (or withdrew consent) before the first scan and 1 additional patient died before the first scan. Thus, the final sample size for responses is n = 46 (T-DM1 only: n = 11; T-DM1 + Palbociclib: n = 35).
Measure: Count of Participants; unit: Participants
Arm/Group | T-DM1 With Palbociclib | Single Agent T-DM1
Number analyzed (Participants) | 35 | 11
Participants
  Overall Response Rate | 15 | 2
  Disease Control Rate | 30 | 7
  Complete Response | 3 | 0
  Partial Response | 12 | 2
  Stable Disease | 15 | 5
  Progressive Disease | 5 | 4

3. Secondary Outcome: Estimate Overall Survival
Description: Estimate overall survival of T-DM1+Palbociclib treatment regimen. Overall survival (OS) is defined as the time from date of first treatment to date of death due to any cause. Patients last known to be alive are censored at their last contact date.
Time Frame: Up to 4 years
Population: We used date of study discontinuation as the censoring date for patients excluded from the survival follow-up file. There are not enough deaths recorded to calculate median OS in the T-DM1 only arm (nor the upper bound of the confidence interval for the T-DM1 + Palbociclib arm).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | T-DM1 With Palbociclib | Single Agent T-DM1
Number analyzed (Participants) | 38 | 14
Months | 35.1 [24.9 to NA] — We used date of study discontinuation as the censoring date for patients excluded from the survival follow-up file. There are not enough deaths recorded to calculate the upper bound of the confidence interval for the T-DM1 + Palbociclib arm. | NA [7.8 to NA] — The upper limit was not reached due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed and collected starting from day 1 of study treatment and continued through the 30 day follow-up period after treatment discontinuation, up to 4 years.
Description: AEs were assessed using the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 for Toxicity and Adverse Event reporting.
  AEs meeting the below criteria were not collected:
  * Hospitalization for elective surgery or routine clinical procedures that are not the result of an AE (e.g., surgical insertion of central line).
  * Disease progression (unless it was attributable by the investigator to the study therapy).
Arm/Group | T-DM1 With Palbociclib | Single Agent T-DM1
All-Cause Mortality (participants affected / at risk) | 5/38 | 4/14
Serious Adverse Events (participants affected / at risk) | 8/38 | 3/14
Other Adverse Events (participants affected / at risk) | 38/38 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DM1 With Palbociclib (N=38) | Single Agent T-DM1 (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DM1 With Palbociclib (N=38) | Single Agent T-DM1 (N=14)
Anaemia (Blood and lymphatic system disorders) | 18 (64) | 4 (10)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Eye disorder (Eye disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 5 (8)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (20) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 12 (16) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (4) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 17 (22) | 8 (9)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 7 (16) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (10) | 5 (7)
Chills (General disorders) | 3 (3) | 2 (2)
Face oedema (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 17 (30) | 7 (9)
Influenza like illness (General disorders) | 3 (3) | 3 (3)
Localised oedema (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (5) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 0 (0)
Pain (General disorders) | 2 (3) | 2 (2)
Pyrexia (General disorders) | 4 (7) | 0 (0)
Corona virus infection (Infections and infestations) | 4 (4) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (8) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 15 (29) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 18 (51) | 7 (11)
Blood alkaline phosphatase increased (Investigations) | 10 (12) | 2 (2)
Blood bilirubin decreased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 7 (12) | 0 (0)
Ejection fraction decreased (Investigations) | 2 (2) | 0 (0)
Haematocrit decreased (Investigations) | 3 (5) | 0 (0)
Lymphocyte count decreased (Investigations) | 16 (50) | 1 (3)
Neutrophil count decreased (Investigations) | 32 (162) | 0 (0)
Neutrophil percentage decreased (Investigations) | 2 (5) | 0 (0)
Platelet count decreased (Investigations) | 29 (178) | 3 (14)
Red blood cell count decreased (Investigations) | 5 (8) | 0 (0)
Red cell distribution width increased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 5 (8) | 2 (3)
White blood cell count decreased (Investigations) | 29 (162) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 9 (11) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (27) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (8) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (23) | 3 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (14) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 17 (19) | 4 (6)
Paraesthesia (Nervous system disorders) | 6 (6) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (9) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (20) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Contusion (Vascular disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 4 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was originally a 2-arm, randomized study (T-DM1 with Palbociclib and single agent T-DM1); however, due to the COVID-19 pandemic restrictions and slow accrual, the study design was updated to a single arm study of T-DM1 with Palbociclib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03530696/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT03530696/ICF_001.pdf